CLINICAL TRIAL: NCT00227019
Title: Phase II Trial of Bevacizumab in Combination With Pemetrexed as Second Line Therapy in Patients With Stable Brain Metastases From Non-small Cell Lung Cancer (NSCLC) (Excluding Squamous Cell Carcinoma)
Brief Title: Phase 2 Trial of Bevacizumab in Combination With Pemetrexed
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heather Wakelee (Other)
Collaborators: Eli Lilly and Company (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Heather Wakelee, Assistant Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-00892; 95913 (Other: Stanford University Alternate IRB Approval Number); LUN0014 (Other: OnCore)
Record Dates: First submitted 2005-09-08; First posted 2005-09-27 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Non-small Cell Lung Cancer (NSCLC); Lung Cancer; Neoplasm Metastasis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasm Metastasis | interventions — Bevacizumab; Pemetrexed; Vitamin B 12; Folic Acid; Leucovorin; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bevacizumab+ pemetrexed (Experimental): pemetrexed (500 mg/m² IV) + bevacizumab (15 mg/kg IV). In addition to Vitamin B12 + Folate + Dexamethasone
  Interventions: Drug: Bevacizumab; Drug: Pemetrexed; Drug: Vitamin B12; Drug: Folate; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bevacizumab — 15 mg/kg, IV over 10 minutes every 3 weeks
  Other Names: Avastin
Drug: Pemetrexed — 500 mg/m²; IV over 10 minutes every 3 weeks
  Other Names: Alimta
Drug: Vitamin B12 — 1000 micrograms, IM injection 1-2 weeks prior to treatment and repeated every 9 weeks until last dose of pemetrexed
  Other Names: cobalamin; Vit B12
Drug: Folate — 350 to 1000 micrograms 1 week prior to treatment and 3 weeks after last pemetrexed dose
  Other Names: folacin; Folic acid; pteroyl-L-glutamic acid; pteroyl-L-glutamate; pteroylmonoglutamic acid; vitamin B9; vitamin Bc
Drug: Dexamethasone — 4 mg; oral, twice a day at the following times: the day before, of and after each dose of pemetrexed
  Other Names: Decadron

SUMMARY:
This trial evaluated the safety of combining bevacizumab and pemetrexed in non-small cell lung cancer (NSCLC) patients with stable brain metastases as second-line chemotherapy, while evaluating progression-free survival (PFS) and overall survival (OS).

DETAILED DESCRIPTION:
Brain metastases are a common complication of advanced non-small-cell lung cancer (NSCLC) both at initial presentation and at the time of disease progression. Patients with brain metastases have often been excluded from large randomized phase III trials due to concerns of poorer survival and impaired ability of drugs to cross the blood-brain barrier. However, as survival has improved, some trials have included such patients, often finding similar benefit to patients with metastatic disease elsewhere.

Bevacizumab is a recombinant, humanized monoclonal antibody against vascular endothelial growth factor, has emerged as an important adjunct to platinum-based chemotherapy doublets for use in advanced NSCLC. This drug is normally used as a first line chemotherapy. Pemetrexed is a multi-targeted anti-folate agent,which is approved for use in first-line (with platinum), maintenance, and second-line treatment of advanced nonsquamous NSCLC. Based on the efficacy of pemetrexed as a second line agent and the safety questions surrounding bevacizumab in those with treated brain metastases, a trial was designed to look at the combination of both agents as a second line therapy in NSCLC patients with treated stable brain metastases

ELIGIBILITY:
Inclusion Criteria:

* Advanced stage NSCLC excluding squamous cell histology with measurable or evaluable disease.
* Stable brain metastases required, no longer requiring active therapy such as steroid medications, which have been previously treated with radiation or surgery or both and have been documented to be stable on repeat imaging done at least one month after completion of therapy.
* Prior therapy with one standard doublet front-line regimen for NSCLC (platinum containing)
* Life expectancy of at least 3 months
* ECOG Performance status 0-1
* Age 18 or higher
* Use of effective means of contraception (men and women) in subjects of child-bearing potential
* Ability/willingness to comply with vitamin supplementation including vitamin B 12 and folic acid started at least 1 week before first dose of pemetrexed and continued for at least 3 weeks after last dose
* Ability/willingness to take dexamethasone the day before, of and after pemetrexed administration
* Drainage of any clinically significant effusion
* Ability to sign informed consent

Exclusion Criteria:

* Treatment with more than one prior chemotherapy regimen (unless one regimen was stopped for toxicity reasons with a different regimen replacement regimen started immediately and patient completed only 4-6 total cycles of first-line treatment. One prior regimen (up to 4 cycles) of neoadjuvant or adjuvant therapy for early stage disease will also be allowed.
* Prior treatment with pemetrexed or bevacizumab
* Prior chemotherapy within 28 days (6 weeks for BCNU, CCNU or mitomycin-C)
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in any other experimental drug study
* Concomitant chemotherapy, radiotherapy or investigational agents
* Uncontrolled effusion (large pleural or peritoneal effusion or small/moderate effusion which requires drainage for symptom management)
* Evidence of bleeding diathesis or coagulopathy
* Use of anti-coagulant agents including warfarin, heparin, aspirin, NSAIDs
* Pregnant (positive pregnancy test) or lactating women
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to day 0
* Urine protein:creatinine ratio greater than or equal to 1.0 at screening
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0
* Serious, non-healing wound, ulcer, or bone fracture
* Lung carcinoma of squamous cell histology or any histology in close proximity to a major vessel, or with significant cavitation as assessed by treating investigator in consultation with an attending radiologist
* History of hemoptysis (bright red blood of 1/2 teaspoon or more)
* Neutrophils < 1.5 x 10^9/ L
* Hemoglobin <10.0 g/dl
* Platelets <100 x 10^9/ L
* Serum glutamic oxaloacetic transaminase (SGOT/ AST) or serum glutamic pyruvic transaminase (SGPT/ ALT) > 2.5 times upper limits of normal
* Creatinine > 1.5 times upper limits of normal
* Significant co-morbidities including:

  * Blood pressure of greater than 150/100 mmHg
  * Unstable angina
  * New York Heart Association (NYHA) Grade II or greater congestive heart failure
  * History of myocardial infarction within 6 months
  * History of stroke within 6 months
  * Clinically significant peripheral vascular disease
* Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-03; Primary Completion 2010-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather A. Wakelee, Principal Investigator — Stanford University
Locations (4):
- United States (4):
  - Stanford University School of Medicine, Stanford, California
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Cooper Cancer Institute, Voorhees Township, New Jersey
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab Plus Pemetrexed: Treatment group is adult patients with metastatic nonsquamous, non-small cell lung cancer (NSCLC) and stable brain metastases after progression on a platinum doublet regimen for advanced disease. All patients received pemetrexed (500 mg/m² IV) + bevacizumab (15 mg/kg IV) every 3 weeks.
Period: Overall Study
Arm/Group | Bevacizumab Plus Pemetrexed
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Adult patients with advanced stage nonsquamous NSCLC and stable treated metastatic disease in the brain were eligible if they were candidates for second-line therapy after progression on a platinum doublet regimen for advanced disease.
Arm/Group | Bevacizumab Plus Pemetrexed
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 60 [33 to 78]
Gender [Count of Participants; unit: Participants]
  Female | 9
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: participants] — ECOG performance status
  * 0 = Fully active, able to carry on all pre-disease performance without restriction
  * 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg, light house work, office work
  * 2 = Unable to work, must sit or lie > 50% waking hours
  * 3 = Capable of limited selfcare; confined to bed or chair > 50% waking hours
  * 4 = Completely disabled; cannot carry on any selfcare; totally confined to bed/chair
  * 5 = Deceased
  participants
    0-1 | 15
    2 | 1
Histology [Number; unit: participants] — Histology refers to the type of non-small cell lung cancer (NSCLC)
  participants
    Adeno-carcinoma | 12
    Large cell carinoma | 0
    Not otherwise specified (NOS) | 4

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Central Nervous System (CNS) Hemorrhagic Events
Description: Number of events of brain or central nervous system (CNS) bleeding
Time Frame: 18 months
Population: All participants in this study are included in the analysis population
Measure: Number; unit: CNS hemorrhagic events
Groups:
- Bevacizumab + Pemetrexed: Treatment group is adult patients with metastatic non squamous, non-small cell lung cancer (NSCLC) and stable brain metastases after progression on a platinum doublet regimen for advanced disease. All patients received pemetrexed (500 mg/m² IV) + bevacizumab (15 mg/kg IV) every 3 weeks.
Arm/Group | Bevacizumab + Pemetrexed
Number analyzed (Participants) | 16
CNS hemorrhagic events | 0

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of documented disease progression or death.
  Kaplan-Meier survival curves for PFS were generated with IBM SPSS Statistics version 19.0 (SPSS, Inc, Chicago, IL).
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Pemetrexed
Number analyzed (Participants) | 16
months | 7.2 [5.5 to 9.0]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is defined as the duration of time from start of treatment to deat.
  Kaplan-Meier survival curves for OS were generated with IBM SPSS Statistics version 19.0 (SPSS, Inc, Chicago, IL).
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bevacizumab + Pemetrexed: Treatment group is adult patients with metastatic nonsquamous, non-small cell lung cancer (NSCLC) and stable brain metastases after progression on a platinum doublet regimen for advanced disease. All patients received pemetrexed (500 mg/m² IV) + bevacizumab (15 mg/kg IV) every 3 weeks.
Arm/Group | Bevacizumab + Pemetrexed
Number analyzed (Participants) | 16
months | 14.8 [9.4 to 21.0]

ADVERSE EVENTS:
Time Frame: 18 Months
Groups:
- Bevacizumab Plus Pemetrexed: Treatment group is adult patients with metastatic non squamous, non-small cell lung cancer (NSCLC) and stable brain metastases after progression on a platinum doublet regimen for advanced disease. All patients received pemetrexed (500 mg/m² IV) + bevacizumab (15 mg/kg IV) every 3 weeks.
Arm/Group | Bevacizumab Plus Pemetrexed
Serious Adverse Events (participants affected / at risk) | 8/16
Other Adverse Events (participants affected / at risk) | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab Plus Pemetrexed (N=16)
Infection (General disorders) | 6
Dyspnea/ respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
Fatigue (General disorders) | 3
Neutropenia +/- fever (Blood and lymphatic system disorders) | 3
Elevated creatinine/ Actue Renal failure (ARF) (Blood and lymphatic system disorders) | 1
Thrombosis/ deep vein thrombosis (DVT) (Blood and lymphatic system disorders) | 2
Confusion (General disorders) | 1
Hyperglycemia (Blood and lymphatic system disorders) | 1
Hyponatremia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Pain (General disorders) | 1
Seizure-like activity (Musculoskeletal and connective tissue disorders) | 1
Syncope (Blood and lymphatic system disorders) | 1
Weight gain (General disorders) | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab Plus Pemetrexed (N=16)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Allergic reaction (Immune system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Anemia (Blood and lymphatic system disorders) | 2
Blurred vision (Eye disorders) | 3
Bruising (Injury, poisoning and procedural complications) | 1
Catheter related infection (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Chills (General disorders) | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 2
Constipation (Gastrointestinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Creatinine increased (Investigations) | 2
Creatinine increased (Metabolism and nutrition disorders) | 8
Anorexia (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Localized edema (General disorders) | 2
Edema limbs (General disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Erectile dysfunction (Reproductive system and breast disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1 — eye irritation
Fatigue (General disorders) | 11
Fever (General disorders) | 2
Gait disturbance (General disorders) | 1
Vascular disorders - Other, specify (Vascular disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 3
Hearing impaired (Ear and labyrinth disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Hot flashes (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Injection site reaction (General disorders) | 1
Insomnia (Psychiatric disorders) | 3
Periodontal disease (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Fever (General disorders) | 3 — Low grade fever
Amnesia (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Neutrophil count decreased (Investigations) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pain (General disorders) | 12
Pancreatitis (Gastrointestinal disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3
Upper respiratory infection (Infections and infestations) | 2
Infections and infestations - Other, specify (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Hepatobiliary disorders - Other, transiminitis (Hepatobiliary disorders) | 1
Tremor (Nervous system disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Weight loss (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No